CLINICAL TRIAL: NCT06102421
Title: Evaluation of the Effectiveness of Extracorporeal Shockwave Therapy in Patients With Patellar Tendinopathy on Its Micromorphology
Status: Completed | Type: Observational
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Stanislav Machač, Ph.D, Principal investigator, University Hospital, Motol
Other Study IDs: EK-980/23
Record Dates: First submitted 2023-10-20; First posted 2023-10-26 (Actual); Results first posted 2025-04-11 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Patellar Tendinopathy
Keywords: Patellar Tendinopathy; Extracorporeal Shock Wave Therapy; Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Symptomatic patellar tendon (patellar tendinopathy) treated by ESWT: The included patients show signs of unilateral patellar tendinopathy and were included in the study in accordance with the inclusion and exclusion parameters. Data of clinical symptoms and morphological measures of symptomatic patellar tendons of enrolled participants are allocated to this group. Participants will receive a low-energy focused ESWT in accordance with study protocol.
  ESWT will be applied 4 times with an interval of 7 days from the BTL-6000 FSWT device with piezoelectric generator. The energy can vary between 0.12-0.20 mJ/mm2 based on the pain toleration, frequency 5 Hz, total number of shocks 2x2000. The application of the first set of shocks will be semi-static at the location of the largest USG defined pathology in the patellar tendon and the second set of shocks will be performed dynamically to the proximal tendon. These parameters were selected in accordance to ISMST guidelines.
  Interventions: Device: BTL-6000 FSWT
- Healthy tendon: The asymptomatic tendons of enrolled patient are allocated to this group and are considered healthy based on clinical and ultrasound examination of the patellar tendon.
  In this group, no specific treatment will be performed, only patellar tendon morphology will be monitored through time.

INTERVENTIONS:
Device: BTL-6000 FSWT — Low-energy focused extracorporeal shockwave therapy will be applied 4 times with an interval of 7 days from the BTL-6000 FSWT device with piezoelectric generator. The energy can vary between 0.12-0.20 mJ/mm2 based on the pain toleration, frequency 5 Hz, total number of shocks 2x2000. The application of the first set of shocks will be semi-static at the location of the largest USG defined pathology in the patellar tendon and the second set of shocks will be performed dynamically to the proximal tendon. These parameters were selected in accordance to ISMST guidelines.
  Groups: Symptomatic patellar tendon (patellar tendinopathy) treated by ESWT

SUMMARY:
This work is designed as a prospective cohort study, in which the effects of low-energy focused extracorporeal shock wave therapy (ESWT) in patients with Patellar tendinopathy (PT) will be monitored on its micromorphology. It is estimated that at least 21 patients will participate. In addition, there will be a small control group of healthy tendons which will be monitored to observe magnitude of natural changes.

DETAILED DESCRIPTION:
This work is designed as a prospective cohort study, in which the effects of low-energy focused extracorporeal shock wave therapy (ESWT) in patients with Patellar tendinopathy (PT) will be monitored on its micromorphology. It is estimated that at least 21 patients will participate. In addition, there will be a small control group of healthy tendons which will be monitored to observe magnitude of natural changes.

The research within one patient will last a total of 16 weeks from the initial to the final examination. Potential participants will be selected based on the recommendation of a specialist doctor and their suitability will be assessed according to the inclusion criteria. They will then be invited to an initial examination. This will include an objective examination by a physiotherapist, a subjective assessment by the patient and an ultrasonographic (USG) examination followed by a micromorphological analysis using special software.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a recreational athlete performing intensive sport activity loading patellar tendon (running, jumping, strength training etc.) at least 3 days in a week for minimum of 1 hour per session,
* is in age between 18-40 years,
* has a patellar tendon pain, which limits (at least in part) the quality of normal daily or sports activities,
* has clinical manifestation of patellar tendinopathy (pain and impaired function) confirmed by clinician,
* has symptoms only in one leg, the other one is asymptomatic.

Exclusion Criteria:

* Any contraindication for ESWT is present (according to International Society for Medical Shockwave Treatment (ISMST) consensus at https://shockwavetherapy.org),
* Patient is aware of any symptomatic mechanical tendon damage in the past (e.g., partial or complete rupture in relation to the injury),
* neurological, oncological, or systemic disease (e.g., neuropathy, lupus or rheumatic arthritis) coexists,
* is/was already treated for PT elsewhere (e.g., platelet-rich plasma therapy, physiotherapy)
* is using blood thinning medications or statins.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The monitored population are patients suffering from symptomatic, unilateral, recently untreated patellar tendinopathy lasting at least 3 months, age between 18 - 40 years. They were not diagnosed with a rheumatic, neurological or oncological disease and have no contraindication for ESWT.
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-02-25 (Actual); Study Completion 2024-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislav Machac, PhD, Study Chair — University Hospital Motol and 2nd Faculty of Medicine, Charles University
Locations (1):
- University Hospital Motol and 2nd Faculty of Medicine, Charles University, Prague, Czechia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Symptomatic Patellar Tendon (Patellar Tendinopathy) Treated by ESWT | Healthy Tendon
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Symptomatic Patellar Tendon (Patellar Tendinopathy) Treated by ESWT | Healthy Tendon | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 21 | 42
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.8 (9.1) | 29.8 (9.1) | 29.8 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 16 | 16 | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Czechia | 21 | 21 | 42
BMI [Mean (Standard Deviation); unit: kg/m2] | 24.2 (3.2) | 24.2 (3.2) | 24.2 (3.2)
Symptom duration [Mean (Standard Deviation); unit: months] | 19.6 (16.1) | 19.6 (16.1) | 19.6 (16.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Peak Spatial Frequency Radius at the Site of Pathology
Description: Measured by spatial frequency analysis software from ultrasound picture in mm. In a linear view with specific settings of ultrasound machine, the site of the largest pathology is selected, then the image is saved and uploaded to the software that evaluates the PSFR parameter.
Time Frame: Change of initial values at 16 weeks follow up after beginning of the therapy.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Symptomatic Patellar Tendon Treated by ESWT - Baseline: Baseline values
  The included patients show signs of unilateral patellar tendinopathy and were included in the study in accordance with the inclusion and exclusion parameters. Data of clinical symptoms and morphological measures of symptomatic patellar tendons of enrolled participants are allocated to this group. Participants will receive a low-energy focused ESWT in accordance with study protocol.
  ESWT will be applied 4 times with an interval of 7 days from the BTL-6000 FSWT device with piezoelectric generator. The energy can vary between 0.12-0.20 mJ/mm2 based on the pain toleration, frequency 5 Hz, total number of shocks 2x2000. The application of the first set of shocks will be semi-static at the location of the largest USG defined pathology in the patellar tendon and the second set of shocks will be performed dynamically to the proximal tendon. These parameters were selected in accordance to ISMST guidelines.
- Symptomatic Patellar Tendon Treated With ESWT - Follow-up: Follow-up values
  The included patients show signs of unilateral patellar tendinopathy and were included in the study in accordance with the inclusion and exclusion parameters. Data of clinical symptoms and morphological measures of symptomatic patellar tendons of enrolled participants are allocated to this group. Participants will receive a low-energy focused ESWT in accordance with study protocol.
  ESWT will be applied 4 times with an interval of 7 days from the BTL-6000 FSWT device with piezoelectric generator. The energy can vary between 0.12-0.20 mJ/mm2 based on the pain toleration, frequency 5 Hz, total number of shocks 2x2000. The application of the first set of shocks will be semi-static at the location of the largest USG defined pathology in the patellar tendon and the second set of shocks will be performed dynamically to the proximal tendon. These parameters were selected in accordance to ISMST guidelines.
Arm/Group | Symptomatic Patellar Tendon Treated by ESWT - Baseline | Symptomatic Patellar Tendon Treated With ESWT - Follow-up
Number analyzed (Participants) | 21 | 21
mm | 2.119 (0.148) | 2.234 (0.133)

2. Primary Outcome: Change in VISA-P Questionnaire Score
Description: The VISA-P questionnaire is standardized questionnaire for patients with Patellar tendinopathy. The results are recorded in points (0-100 points). The higher score indicates patients better condition.
Time Frame: Change of initial values at 16 weeks follow up after beginning of the therapy.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Symptomatic Patellar Tendon Treated by ESWT - Baseline: Baseline values.
  The included patients show signs of unilateral patellar tendinopathy and were included in the study in accordance with the inclusion and exclusion parameters. Data of clinical symptoms and morphological measures of symptomatic patellar tendons of enrolled participants are allocated to this group. Participants will receive a low-energy focused ESWT in accordance with study protocol.
  ESWT will be applied 4 times with an interval of 7 days from the BTL-6000 FSWT device with piezoelectric generator. The energy can vary between 0.12-0.20 mJ/mm2 based on the pain toleration, frequency 5 Hz, total number of shocks 2x2000. The application of the first set of shocks will be semi-static at the location of the largest USG defined pathology in the patellar tendon and the second set of shocks will be performed dynamically to the proximal tendon. These parameters were selected in accordance to ISMST guidelines.
- Symptomatic Patellar Tendon Treated by ESWT - Follow-up: Follow-up values.
  The included patients show signs of unilateral patellar tendinopathy and were included in the study in accordance with the inclusion and exclusion parameters. Data of clinical symptoms and morphological measures of symptomatic patellar tendons of enrolled participants are allocated to this group. Participants will receive a low-energy focused ESWT in accordance with study protocol.
  ESWT will be applied 4 times with an interval of 7 days from the BTL-6000 FSWT device with piezoelectric generator. The energy can vary between 0.12-0.20 mJ/mm2 based on the pain toleration, frequency 5 Hz, total number of shocks 2x2000. The application of the first set of shocks will be semi-static at the location of the largest USG defined pathology in the patellar tendon and the second set of shocks will be performed dynamically to the proximal tendon. These parameters were selected in accordance to ISMST guidelines.
Arm/Group | Symptomatic Patellar Tendon Treated by ESWT - Baseline | Symptomatic Patellar Tendon Treated by ESWT - Follow-up
Number analyzed (Participants) | 21 | 21
score on a scale | 68.4 (8.2) | 83.3 (7.1)

3. Primary Outcome: Change in P6 Parameter at the Site of Pathology
Description: Measured by spatial frequency analysis software from ultrasound picture in mm. In a linear view with specific settings of ultrasound machine, the site of the largest pathology is selected, then the image is saved and uploaded to the software that evaluates the P6 parameter.
Time Frame: Change of initial values at 16 weeks follow up after beginning of the therapy.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Symptomatic Patellar Tendon Treated With ESWT - Baseline: Baseline values
  The included patients show signs of unilateral patellar tendinopathy and were included in the study in accordance with the inclusion and exclusion parameters. Data of clinical symptoms and morphological measures of symptomatic patellar tendons of enrolled participants are allocated to this group. Participants will receive a low-energy focused ESWT in accordance with study protocol.
  ESWT will be applied 4 times with an interval of 7 days from the BTL-6000 FSWT device with piezoelectric generator. The energy can vary between 0.12-0.20 mJ/mm2 based on the pain toleration, frequency 5 Hz, total number of shocks 2x2000. The application of the first set of shocks will be semi-static at the location of the largest USG defined pathology in the patellar tendon and the second set of shocks will be performed dynamically to the proximal tendon. These parameters were selected in accordance to ISMST guidelines.
Arm/Group | Symptomatic Patellar Tendon Treated With ESWT - Baseline | Symptomatic Patellar Tendon Treated With ESWT - Follow-up
Number analyzed (Participants) | 21 | 21
mm | 1.119 (0.022) | 1.099 (0.022)

4. Secondary Outcome: Change in Tendon Diameter at the Place of Maximum Tendon Width
Description: Measured by tools in ultrasound machine in mm. In linear view is selected maximal width place, then the tendon diameter is measured using device tools.
Time Frame: Change of initial values at 16 weeks follow up after beginning of the therapy.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Symptomatic Patellar Tendon Treated by ESWT - Baseline | Symptomatic Patellar Tendon Treated by ESWT - Follow-up
Number analyzed (Participants) | 21 | 21
mm | 4.87 (0.74) | 4.40 (0.73)

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: No adverse effects (serious or others) were reported during treatment, after treatment and also during follow-up period.
Arm/Group | Symptomatic Patellar Tendon (Patellar Tendinopathy) Treated by ESWT | Healthy Tendon
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-04): https://cdn.clinicaltrials.gov/large-docs/21/NCT06102421/Prot_SAP_000.pdf